CLINICAL TRIAL: NCT04485312
Title: Chance to Avoid New Caries by Adding Chlorhexidine Containing Chemotherapeutic Agent to the Conventional Preventive Protocol for Patients With Special Needs
Brief Title: Chance to Avoid New Caries by Adding Chlorhexidine to the Preventive Protocol in Adolescent Special Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Katreen Tawfik, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: abcxyz
Record Dates: First submitted 2020-07-18; First posted 2020-07-24 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Disabilities Multiple

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caries preventive protocol (Active Comparator): preventive protocol for special needs ( tooth brushing , topical fluoride and mouth wash)
  Interventions: Behavioral: preventive protocol
- chlorhexidine varnish added to the caries preventive protocol (Other): chlorhexidine varnish preventive caries protocol for special needs
  Interventions: Behavioral: chlorhexidine added to the preventive protocol

INTERVENTIONS:
Behavioral: preventive protocol — preventive protocol
  Arms: caries preventive protocol
Behavioral: chlorhexidine added to the preventive protocol — chlorhexidine varnish added to the preventive protocol
  Arms: chlorhexidine varnish added to the caries preventive protocol

SUMMARY:
Adolescent Special need individuals are most need of easy forms of antibacterial agents, so in this study, using chemotherapeutic agents like the newly introduced varnish containing chlorhexidine seems to be a quite promising tool for local delivery to patients with special needs . Chlorhexidine is a wide spectrum very effective bactericidal used for years against the oral flora while fluorides are well known with their antibacterial ability. This may be an excellent way to reduce the risk assessment in adolescent special needs patients.

DETAILED DESCRIPTION:
Participants will be divided into two groups according to the tested regimen, where (A1) represents participants exposed to risk based conventional protocol, (A2) represents participants exposed to chlorhexidine containing varnish and risk based conventional preventive protocol. The study will be carried over a period of 10 months (one academic year), the study will be divided into three phases Phase I: Information of the Cariogram parameters (caries experience, diet content, diet frequency, plaque amount, mutans streptococci, fluoride program, saliva secretion and saliva buffer capacity) will be collected, which will be used to generate the individual caries profile, based on which the participants will be divided into 2 risks groups. Phase II: Risk based preventive program will be implemented including the restorative part. Phase III: At the end of 10 months, caries profile will be generated again

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of disability like : autism and down syndrome.
* Must be able to open his/her mouth for varnish application

Exclusion Criteria:

* systemically unhealthy patients with fetal diseases
* Age below 13 and above 18

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
chance to avoid new caries | 10 months
  % of the green sector in the cariogram

CONTACTS AND LOCATIONS:
Overall Officials: katreen tawfik, master, Principal Investigator — cairo U
Locations (1):
- School, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
publications in journal
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year
Access Criteria: online access